CLINICAL TRIAL: NCT05876429
Title: Optimizing the Safety of Inter-Hospital Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Crico (Other)
Responsible Party: Principal Investigator, Stephanie Mueller, Associate Physician, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020P001945
Record Dates: First submitted 2023-04-06; First posted 2023-05-25 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Inpatient Facililty Diagnoses

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Intervention: Current Transfer Process (Active Comparator): Control: Transfer patients are admitted per usual based on existing processes for GMS, Cardiology, and Oncology services. Data collection assesses clinician reported feedback on the logistics for each patient transfer, and issues along the transfer supply chain.
  Interventions: Other: Existing Transfer Patient Admission Process
- Post-Intervention: Implementing Standardized Accept Note (Experimental): Intervention Arm: After engaging stakeholders and finalizing a standardized accept note for transfer patients, appropriate staff will be trained on the use of the note and the note will be implemented in the transfer patient admission process. Data collection will assess clinician reported feedback on the logistics for each patient transfer, and issues along the transfer supply chain, post-intervention.
  Interventions: Other: New Standardized Accept Note

INTERVENTIONS:
Other: New Standardized Accept Note — A standardized accept note for transfer patients will be implemented, after stakeholder engagement and subsequent finalization.
  Arms: Post-Intervention: Implementing Standardized Accept Note
Other: Existing Transfer Patient Admission Process — Maintain existing transfer patient admission processes, across GMS, Cardiology, and Oncology services.
  Arms: Pre-Intervention: Current Transfer Process

SUMMARY:
This proposal aims to design, implement and rigorously evaluate a standardized accept note in a population of patients that have high frequency of IHT, including patients transferred to the general medical (GMS), cardiology and oncology services at a large tertiary care hospital. This study will improve scientific knowledge by quantifying the patient safety impact of an intervention to improve communication of essential clinical information during IHT. If shown effective, the results of this study can be used to improve clinical practice by establishing evidence-based communication guidelines for broad dissemination. We will also establish technical feasibility by successfully implementing this tool within our EHR (Epic, Verona, WI), allowing for feasible adoption and dissemination to other institutions with similar EHR capabilities. Lastly, we will address malpractice risk by investigating a strategic intervention aimed at reducing known contributors to patient harm during IHT, a high-risk transition in care that involves transfer of high-acuity patients between providers, settings and systems of care.

DETAILED DESCRIPTION:
Inter-hospital transfer (IHT), commonly performed to provide patients with more specialized care, involves transfer of patients between providers, settings and systems of care, leaving these patients vulnerable to the risks of discontinuity of care. Standardized communication tools, which have been successful at reducing patient harm among other similar hospital-based care transitions (i.e., intra-hospital patient handoffs), have been under-utilized during IHT to-date, leaving the process largely non-standardized and variable.

The overall goal of this proposal is to optimize patient safety during IHT to GMS, cardiology and oncology services, collectively comprising nearly 50% of all IHT to Brigham and Women's Hospital (BWH), by leveraging our pilot work to design, implement and rigorously evaluate a standardized communication tool to be used during IHT. We propose the following Specific Aims to accomplish this goal:

Aim 1. Utilize pilot data and stakeholder input to revise the standardized accept note.

Aim 2a. Implement the revised standardized accept note for all patients transferred from another acute care hospital to the GMS, cardiology, and oncology inpatient services at BWH.

Aim 2b. Shift the responsibility of documentation of the accept note from a diffuse group of individual clinicians to a small group of dedicated nurses within the Access Center.

Aim 3. Prospectively evaluate the impact of the intervention on patient safety outcomes, including: clinician-reported medical errors and adverse events, length of stay after transfer, rapid-response or code within 6-hours of transfer, ICU-transfer within 24-hours of transfer, and 3-day and in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* source of admission is inpatient transfer from another acute care hospital
* admitted to general medical service
* admitted to cardiology service
* admitted to oncology service
* admitted to ICU service
* age >= 18

Exclusion Criteria:

* source of admission is other than inpatient transfer
* admitted to service other than listed above
* age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1658 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
clinician-reported medical errors and adverse events | Up to 2 weeks
  Medical errors and adverse events measured as the total number of medical errors per patient

SECONDARY OUTCOMES:
Presence of any adverse event after transfer | up to 2 weeks
  Clinician reported adverse events for each transferred patient
Preventable adverse event after transfer | up to 2 weeks
Ameliorable adverse event after transfer | up to 2 weeks
Length of stay of hospitalization after transfer | up to 2 weeks
ICU-transfer within 24 hours of transfer | Up to 24 hours
In-hospital mortality | up to 30 weeks
presence of accept note | Up to 24 hours
timeliness of accept note | Up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Mueller, M.D., M.P.H., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT05876429/Prot_000.pdf